CLINICAL TRIAL: NCT05888428
Title: Regulatory Clearance of a Rehabilitation System for Individuals With Upper Limb Loss
Brief Title: Study of Efficacy of the MyoTrain System in a Population of Individuals With Trans-radial Limb Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Infinite Biomedical Technologies (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Johns Hopkins University (Other); Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Principal Investigator, Rahul Kaliki, Chief Executive Officer, Infinite Biomedical Technologies
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: U44NS119842 (NIH)
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Amputation; Upper Limb
Keywords: amputation; upper limb; myoelectric; training; prosthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Experimental (Experimental): Participants will be provided with the take-home MyoTrain system, which includes the MyoTrain armband, iPad, and MyoTrain software. Participants will progress through the training modules of the MyoTrain software, starting with eliciting paired single DoF antagonistic movements and ending with the proportional control of complex, 2-DoF hand and wrist movements.
  Interventions: Device: MyoTrain
- Control (Active Comparator): Participants will be provided motor imagery exercises that involve brief attempts to move the missing limb in a similar manner to how they would control their pattern recognition system to strengthen their muscles. These exercises do not involve any real-time control feedback.
  Interventions: Behavioral: Motor Imagery

INTERVENTIONS:
Device: MyoTrain — MyoTrain is a virtual prosthesis control training system. From a hardware perspective it consists of an Apple iPad tablet computer and an eight-channel EMG armband, based on the Element electrode platform, which interfaces with the tablet via Bluetooth™. From a software perspective, MyoTrain was developed in the cross-platform Unity 4.0 game development environment.
  Arms: Experimental
Behavioral: Motor Imagery — Motor imagery describes the process by which a prosthesis user mentally simulates the execution of a desired limb movement and activates the musculature of the residual limb that would generate the desired movement.
  Arms: Control

SUMMARY:
The investigators propose to evaluate the efficacy of MyoTrain in a prospective clinical study involving 16 individuals with trans-radial upper-limb loss over a period of 206 days. These individuals will be randomized to Group A (Control Group using standard motor imagery training) and Group B (who are provided the MyoTrain system).

The investigators will test three hypotheses:

1. The use of MyoTrain results in skills transference to control of the final prosthesis
2. The virtual outcome measures in MyoTrain are correlated with real-world functional outcome measures
3. The use of MyoTrain results in improved clinical outcomes as measured by functional, subjective and usage metrics

Following a baseline functional assessment, participants will undergo a 30-day pre-prosthetic training period specific to their assigned Group. After this training period, participants will receive their prosthetic device and occupational therapy consistent with the current clinical care standard, after which they will again undergo clinical assessment. Post-device delivery, participants will then complete 3 56-day blocks of at-home prosthesis use, in between which they will return to clinic for assessment.

ELIGIBILITY:
Inclusion Criteria:

* Trans-radial unilateral limb loss
* Candidate for a 2+ degree-of-freedom myoelectric pattern recognition prosthesis as determined by prosthetist
* Fluent in English
* Age of 18 years or greater

Exclusion Criteria:

* Prior experience with pattern recognition control
* Patients with a residual limb that is unhealed from the amputation surgery
* Patients with easily damaged or sensitive skin who would not tolerate EMG electrodes
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impactive full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean Prosthesis Wear Duration | Days 35-206
  Investigators will measure the mean duration of daily prosthesis wear as a proxy for improved prosthesis acceptance. Prosthesis wear time is defined as the time from when participants dons their prostheses to the time they doff their prostheses. The time points are detected by skin-electrode impedance measurements through the EMG electrodes.

SECONDARY OUTCOMES:
Assessment of Capacity for Myoelectric Control (ACMC) | Days 31, 35, 93, 149, and 206
  In contrast to other instruments, the ACMC does not require a specific set of tools or tasks. Instead, the proctor for the measure chooses an everyday activity, such as setting up a table for snacks or replanting a flower, that is relevant to the study population. As the participants perform the chosen task, a trained rater will assess their capacity for control of their myoelectric prosthesis as represented by 30 items reflecting 6 aspects of quality of myoelectric control. These 6 aspects are "the need for external support," "grip force and opening width," "coordination of both hands, "in different positions and in motion (timing)," "repetitive grip and release," and "the need for visual feedback." Each item is scored on a 4-point scale and converted into linear measures of myoelectric control using Rasch analysis methods on the ACMC website. This outcome measure permits evaluation of bimanual tasks as well as different planes and work spaces of prosthesis use.
Clothespin Relocation Test (CRT) | Days 31, 35, 93, 149, and 206
  The CRT has been adapted from an arm training tool to create an instrument to measure hand function. The CRT is a timed task that measures the time taken to move three standard clothespins from three locations on a horizontal bar to a vertical bar. It tests at least two motor functions simultaneously: hand open/close and wrist pronation/supination.
Module 2 of MyoTrain | Days 0, 31, 35, 93, 149, and 206
  At the onset of the task, a virtual hand is displayed, and a target appears in a location or orientation indicating the final target posture. The targets were specifically designed through iterative focus group testing to ensure they minimally occluded the hand and wrist position during the task. For hand grasp tasks, a translucent grey sphere represents the target location and a red sphere represents a marker tracking the virtual hand's finger position. For wrist pronation/supination tasks, a translucent grey bar appears in a target orientation and a red bar acts a visual marker indicating the virtual hand's current orientation. The goal of the task is to match the hand or wrist orientation with the target location or orientation, respectively. Four metrics are all measured during each task: Movement Completion Rate, Movement Completion Time, Number of Overshoots, and Path Efficiency. The task is failed if the participant does not complete the task within 10 seconds.
Patient-Reported Outcomes Measurement Information System (PROMIS) | Days 0, 31, 35, 93, 149, and 206
  PROMIS is a set of self-reported person-centered measures that evaluate and monitor physical, mental, and social health in adults and children developed by the National Institutes of Health (NIH) to improve outcome reporting across medical sciences. The PROMIS measures were designed to reduce administration time of patient reported outcomes through the use of algorithmically selected surveys. There are 5 instruments of PROMIS that we plan to use for this study: Social Isolation, Ability to Participate, Upper Limb Functionality, Physical Function, and Satisfaction Roles Activities. PROMIS measures are scored according a common metric called the T-score. Typically, the mean of 50 (standard deviation of 10) corresponds to the mean in normative U.S. population.
Daily Mean Number of Movement Bouts | Days 35-206
  The controller does not send any outputs to the prosthesis when "rest" is decoded by the pattern recognition classifier. For all other pattern recognition outputs, movement commands are sent to the prosthesis. Thus, the controller is in a good position to be able to record the amount of prosthesis usage as measured by the frequency of control signals. Such activity is measured in terms of series of continuous movement commands called "movement bouts." The number movement bouts will be recorded and stored in the controller memory.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanger Clinic - Grand Rapids, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No